CLINICAL TRIAL: NCT03280953
Title: Finding the Cut-off Value of Pulse Wave Transit Time (PWTT) to Estimate the Fluid Responsibility
Brief Title: Assessing Fluid Responsiveness With PWTT
Status: Completed | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Gunther Pestel MD, PhD, Consultant of Anesthesiology, Johannes Gutenberg University Mainz
Other Study IDs: 837.004.16
Record Dates: First submitted 2017-04-25; First posted 2017-09-13 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Fluid Therapy; Monitoring, Intraoperative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Assessing fluid responsiveness by PWTT value — PWTT value will be analysed to find the cutoff values compared by esophageal doppler and pulse pressure variation.

SUMMARY:
Pulse wave Transit time (PWTT) is a parameter calculated from ECG and pulseoximeter. It is supposed to help assessing the preload Status and guide intraoperative fluid therapy. This Project aims to validate the benefit of PWTT assessment in an observational clinical fluid study. In case of hypovolemia, patients will receive a fluid Bolus and hemodynamic data from clinical Standard Monitoring, esophageal doppler and PWTT will be recorded before and after the fluid Bolus. Receiver operating characteristic (ROC) curve will be used to determine the validity of PWTT as indicator for fluid responsiveness and its cut off value.

DETAILED DESCRIPTION:
PWTT is determined by measuring the beginning and the end of pulse wave duration and can be calculated as the time interval from the ECG R-wave peak to the rise point of the pulse oximeter wave.

it consists of two components: pre ejection period (PEP) and arterial pulse wave transit time (a-PWTT). PEP is defined as the time from the ECG R wave to the rise point of the aortic root pressure wave. a-PWTT is defined as the time from the rise point of the aortic pressure wave to the rise point of the pulse oximeter wave. a-PWTT is the component which is directly related to the velocity of the pulse wave. However noninvasively, we can measure only PWTT, which also includes PEP. In general, PEP change over short periods of time is negligible in most cases, so we can assume that PWTT corresponds to

a-PWTT. In studies using several studies using animals and healthy volunteers, PWTT showed good correlation with stroke volume or systolic blood pressure. Also in experimental and clinical setting, it is shown that PEP changes indicate change in preloads.

It is not known at this moment, which of the following factors to be considered in processing raw data to acquire accurate PWTT value on predicting fluid responsiveness.

1. The beginning of pulse wave can be assessed by the appearance of either Q wave, which represents the initial phase of depolarisation going through the interventricular septum or R wave, which represents the ventricular depolarisation in ECG.
2. The end of pulse wave duration can be assessed by peripheral plethysmography mostly from a finger tip but also from an ear lobe.
3. The pulse wave time can be simply measured as it is, but can also be adjusted by heart rate using Bazett-Formula.
4. Not only the simple PWTT but also ventilatory induced fluctuation of PWTT (ΔPWTT) may be used for predicting fluid responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 - 80 years old
* elective open abdominal surgery
* clinical indication for direct arterial blood pressure Monitoring
* supine Position intraoperatively

Exclusion Criteria:

* under 18 years, over 80 years old
* pregnant
* no informed consent
* systemic inflammatory response syndrome (SIRS) or Sepsis
* Severe cardiac, coronary or vascular disease
* Arrythmia
* Cardiac valves anomaly
* BMI > 35
* American Society of Anesthesiologists (ASA) physical status classification system: 4
* Lung disease that excludes Ventilation with a tidal volume >8ml/kg
* esophageal pathology
* planned prone position surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled for elective open abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
PWTT change before and after fluid bolus | 1 day
  PWTT recorded before and 1 minute after fluid bolus of 7ml/kg intraoperatively. PWTT values will be calculated: defining PWTT start by either Q-wave or R-wave, defining PWTT end at arrival of the plethysmographic signal either at the finger tip or at the ear lobe, defining PWTT length by either simple measurement or adjusted by the Bazett-Formula. Additionally, as a dynamic parameter respiratory variation of PWTT (ΔPWTT) will be computed.

SECONDARY OUTCOMES:
Heart rate before and after fluid bolus | 1 day
  Heart rate (in beats per minute), derived from intraoperative standard monitoring. This hemodynamic parameter will be measured before and 1min after fluid bolus.
Blood pressure before and after fluid bolus | 1 day
  Systolic blood pressure/diastolic blood pressure/mean arterial pressure (in millimeters of mercury), derived from intraoperative standard monitoring. This hemodynamic parameter will be measured before and 1min after fluid bolus.
Flow Time corrected before and after fluid bolus | 1 day
  Flow Time corrected (in milliseconds) measured by esophageal doppler. This hemodynamic parameter will be measured before and 1min after fluid bolus.
Stroke volume before and after fluid bolus | 1 day
  Stroke volume (in milliliters per heartbeat) measured by esophageal doppler. This hemodynamic parameter will be measured before and 1min after fluid bolus.
Pulse Pressure Variation before and after fluid bolus | 1 day
  Pulse Pressure Variation (as percentage) assessed using arterial pressure monitoring. This hemodynamic parameter will be measured before and 1min after fluid bolus.

CONTACTS AND LOCATIONS:
Overall Officials: Kimiko Fukui-Dunkel, M.D., Ph.D., Principal Investigator — University Medical Center of Johannes Gutenberg University
Locations (1):
- University Medical Center of Johannes Gutenberg University, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rhodes A, Cecconi M, Hamilton M, Poloniecki J, Woods J, Boyd O, Bennett D, Grounds RM. Goal-directed therapy in high-risk surgical patients: a 15-year follow-up study. Intensive Care Med. 2010 Aug;36(8):1327-32. doi: 10.1007/s00134-010-1869-6. Epub 2010 Apr 8. PMID 20376431